CLINICAL TRIAL: NCT03159169
Title: Treatment of Neck and Upper (NU) Limb Pain Using BurstDR Stimulation
Brief Title: Treatment of Neck and Upper Limb Pain Using BurstDR (De Ridder) Stimulation
Acronym: NU-BURST
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The study was discontinued early due to poor recruitment (low enrollment rate)
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SJM-CIP-10194
Record Dates: First submitted 2017-05-11; First posted 2017-05-18 (Actual); Last update posted 2024-09-23 (Actual); Status verified 2024-09

CONDITIONS: Neck Pain; Upper Limb Pain
Keywords: Neck Pain; Upper Limb Pain
MeSH Terms: conditions — Neck Pain | interventions — Spinal Cord Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- study patients (Experimental): Single arm study. Patients will receive Spinal Cord Stimulation (SCS) according to standard clinical procedures.
  Interventions: Device: Spinal Cord Stimulation (SCS)

INTERVENTIONS:
Device: Spinal Cord Stimulation (SCS) — Implantation of SCS electrodes and stimulator according to clinical standards

SUMMARY:
This is a prospective, open label, multicenter feasibility study to evaluate the safety and therapeutic efficacy of BurstDRTM SCS in treating chronic neck pain with or without radiation down to arm/shoulder/upper back

DETAILED DESCRIPTION:
Subjects diagnosed with chronic intractable neck pain with or without radiation down to arm/shoulder/upper back will be considered for inclusion in this study. After baseline evaluation, subjects will undergo a SCS trial using the Abbott Invisible Trial system. At the end of the SCS trial, subjects experiencing at least 50% pain relief, according to average neck VAS (calculated by the average of last 3 days on the pain diary), will be considered for permanent implant and further participation in the study. Pain intensity, quality of life, disability, headache severity, sleep quality, patient satisfaction, anxiety, depression, stimulation sensation and medication usage assessments will be performed at baseline, after SCS trial and at the 3, 6 and 12 month follow up visits.

ELIGIBILITY:
Inclusion Criteria:

* Subject is able to provide informed consent to participate in the study;
* Subject is 18 years of age or older;
* Subject has failed to respond to at least 6 months of conventional treatment which may include pharmacological treatment, physical therapy, and injections;
* Subject has failed to respond to medial branch blocks;
* Subject diagnosed with chronic predominant intractable neck pain with or without radiation down to arm/shoulder/upper back;
* Subject has neck pain intensity of at least 6.0 cm out of 10.0 cm on the average neck pain VAS at baseline (according to the last 3 days of the baseline pain diary);
* Subject is on stable pain medications with a total opioid equivalent of120 mg or less for at least 28 days prior to enrolling in this study, and is willing to stay on those medications with no dose increase until activation of the permanently implanted SCS device;
* Subject's medical record has been evaluated by the Investigator to ensure that the subject is a good candidate for a neurostimulation system;
* Subject is willing to cooperate with the study requirements including compliance with the regimen and completion of all office visits;
* Female candidates of child-bearing potential agree to commit to the use of an effective method of contraception (including but not limited to sterilization, barrier devices, oral contraceptives, intrauterine devices (IUDs), condoms, rhythm method, or abstinence) for the duration of the study

Exclusion Criteria:

* Subject has a current diagnosis of a coagulation disorder, bleeding diathesis, progressive peripheral vascular disease, moderate or severe cervical stenosis determined by existing or new MRI scan performed as part of standard of care, mechanical neck pain originating from cervical facet joint syndrome, post-herpetic neuralgia, spondylolisthesis, retrolisthesis, CRPS (Chronic Regional Pain Syndrome) or uncontrolled diabetes mellitus;
* Subject with significant scoliosis even if surgically corrected;
* Subject is currently participating in a clinical investigation that includes an active treatment arm;
* Subject has been implanted with or participated in a trial period for a neurostimulation system;
* Subject has an infusion pump;
* Subject has evidence of an active disruptive psychological or psychiatric disorder as determined as per standard of care;
* Subject has a current diagnosis of a progressive neurological disease as determined by the Investigator;
* Subject is immunocompromised;
* Subject has an existing medical condition that is likely to require repetitive MRI evaluation in the future (i.e. epilepsy, stroke, multiple sclerosis, acoustic neuroma, tumor);
* Subject has history of cancer requiring active treatment in the last 12 months;
* Subject has an existing medical condition that is likely to require the use of diathermy in the future;
* Subject has documented history of allergic response to titanium or silicone;
* Subject has a documented history of substance abuse (narcotics, alcohol, etc.) or substance dependency in the 6 months prior to baseline data collection;
* Subject is a female candidates of child bearing potential that are pregnant (confirmed by positive urine/blood pregnancy test);
* Subject has life expectancy of less than 1 year;
* Subject is involved in an injury claim under current litigation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2018-05-15 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2022-08-31 (Actual)

PRIMARY OUTCOMES:
Evaluate the change in pain intensity between baseline, trial and long-term follow up evaluations using Visual Analog Scale (VAS) assessments. | 3, 6 and 12 months
  Golden standard self-evaluation of pain intensity

CONTACTS AND LOCATIONS:
Overall Officials: Adnan Al-Kaisy, MD, Principal Investigator — Guy's St. Thomas
Locations (3):
- United Kingdom (3):
  - Southmead hospital, Bristol
  - Guy's St. Thomas Hospital, London
  - University Hospital Southampton NHS Foundation Trust, Southampton

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Al-Kaisy A, Vajramani G, Love-Jones S, Patel NK, Royds J, Palmisani S, Pang D, Wesley S, Park HJ, Raza A, Agnesi F. Multicentre, clinical trial of burst spinal cord stimulation for neck and upper limb pain NU-BURST: a trial protocol. Neurol Sci. 2021 Aug;42(8):3285-3296. doi: 10.1007/s10072-020-04907-3. Epub 2021 Jan 2. PMID 33387056